CLINICAL TRIAL: NCT07408011
Title: Interest of Cryotherapy in Reducing Pain During Radial Arterial Blood Sampling
Acronym: HOURRA
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 29BRC23.0052
Record Dates: First submitted 2026-01-12; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Chronic Respiratory Diseases
Keywords: Arterial blood gas; Pain; Cryotherapy
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Three arms will be compared using a factorial analysis. First, the intervention group (cryotherapy) will be compared with the placebo cream.
  Second, if a significant difference is observed for the primary objective, the lidocaine group will be compared with the placebo cream.
  Third, if a significant difference is observed for the second objective, the lidocaine group will be compared with the intervention group (cryotherapy).
Masking Description: This is an open-label study whose primary objective is to compare cryotherapy with placebo cream for pain. However, both the investigator and the patient will be blinded to whether the applied cream is neutral (placebo) or active (lidocaine), making the comparison between lidocaine and placebo double-blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cryotherapy (Experimental): Application of a medical ice pack on the arm prior to the arterial blood gas procedure
  Interventions: Device: Apllication of medical device ice pack
- Placebo cream (Placebo Comparator): Application of placebo cream on the arm prior the arterial blood gas procedure
  Interventions: Drug: Apllication of cream
- Anesthetic cream (Active Comparator): Application of lidocaine cream on the arm prior arterial blood gas procedure
  Interventions: Drug: Apllication of cream

INTERVENTIONS:
Device: Apllication of medical device ice pack — Application of a medical device pack during 3 minutes on the area where the arterial blood gas will be performed.
  Arms: Cryotherapy
Drug: Apllication of cream — Application of a cream 120 min before on the area where the arterial blood gas will be performed.
  Arms: Anesthetic cream; Placebo cream

SUMMARY:
Arterial puncture for blood gas analysis is a diagnostic procedure used to assess arterial blood gases and monitor a patient's oxygenation status. It is widely regarded by nursing staff as one of the most painful routine procedures. Despite this, the use of local anesthesia prior to arterial puncture remains uncommon in clinical practice.

Several types of anesthetic agents and administration techniques have been evaluated, with mixed results regarding their effectiveness in reducing patient-reported pain. Studies comparing subcutaneous lidocaine injection or ethyl chloride spray to no analgesic intervention have shown that ethyl chloride does not significantly reduce pain. Moreover, the discomfort caused by lidocaine injection appears to be comparable to that of the arterial puncture itself, suggesting limited overall benefit from this approach.

Other investigations have similarly reported a lack of significant pain reduction with ethyl chloride spray, although some contradictory findings exist. Ultrasound-guided arterial puncture has been shown to improve success rates and shorten procedure duration; however, it does not appear to influence pain perception.

The impact of needle size on pain intensity has also been explored, with conflicting results. Some studies found no significant difference in pain when using different gauge needles, while others reported reduced pain with the use of finer needles, such as insulin needles, compared to standard arterial puncture needles.

Topical anesthetic creams combining lidocaine and prilocaine have been assessed in randomized, double-blind trials. These studies found no significant difference between anesthetic and placebo groups in terms of pain intensity or the proportion of painful procedures.

More recently, cryotherapy has been investigated as a non-pharmacological method to reduce pain prior to arterial puncture. Several randomized controlled trials using varying cryotherapy protocols have generally reported a significant reduction in pain compared to control groups, with longer application times appearing to enhance effectiveness.

However, these findings must be interpreted with caution due to methodological limitations. In some studies, sample size calculations were not justified, randomization procedures were poorly described, and reported pain levels were unusually high compared to those typically observed in European populations, raising concerns about external validity. In certain cases, although pain reduction was statistically significant, it did not reach the minimal clinically important difference, limiting its clinical relevance.

Conversely, other trials reported very low pain scores following cryotherapy, suggesting a substantial clinical benefit. The short application time required for cryotherapy also makes it far more practical than topical anesthetic creams, which require prolonged application. This practicality supports its use in both emergency and outpatient settings.

Some authors have noted that blinding is challenging when using cryotherapy and have suggested incorporating placebo interventions in future studies to improve methodological rigor.

Overall, systematic analyses indicate that cryotherapy appears to be a safe and potentially effective method for reducing pain during arterial puncture. Nevertheless, the existing evidence is limited by a high risk of bias, underscoring the need for further high-quality randomized controlled trials.

Conclusion: Given the promising but methodologically constrained evidence, there is a strong justification for conducting a rigorously designed, placebo-controlled randomized trial to accurately assess the effectiveness of cryotherapy in reducing pain associated with radial arterial puncture.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a respiratory condition requiring arterial blood gas sampling via radial puncture
* Patients able to assess their pain using a numerical rating scale
* Patients reporting a pain score of 0 on the numerical scale at the wrist prior to sampling
* Patients with no contraindications or allergies to local anesthetics such as lidocaine/prilocaine
* Patients aged 18 years or older
* Patients affiliated with or benefiting from a social security scheme
* Patients able to give consent and who have signed an informed consent form

Exclusion Criteria:

* Patients reporting a pain score >0 on the numerical rating scale before sampling
* Emergency context requiring immediate arterial blood gas results
* Patients for whom radial arterial puncture is not feasible
* Known hypersensitivity to local amide-type anesthetics or any component of the lidocaine/prilocaine cream
* Pregnant or breastfeeding women
* Refusal to participate
* Patients under legal guardianship or conservatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2029-11-01 (Estimated)

PRIMARY OUTCOMES:
pain, measured on a 0-10 numerical rating scale | At inclusion
  Pain will be measured with the 0-10 numerical rating scale : 0 = no pain, and 10 = the worse pain

SECONDARY OUTCOMES:
the pain , measured with the 0-10 numerical rating scale experienced during the puncture (between the use of a cream combining two local anesthetics (lidocaine/prilocaine) and a placebo cream) | At inclusion
  the pain will be measured with the 0-10 numerical rating scale: 0 = no pain, and 10 = the worse pain
Compare heart rate before the procedure between groups | Before Procedure
  the heart rate will be measured with a pulse oxymeter
Compare heart rate during the procedure between groups | during Procedure
  heart rate will be measured during the procedure with a pulse- oxymeter
Compare heart rate after the procedure between groups | after Procedure
  heart rate will be measured at the end of the procedure with a pulse- oxymeter
Compare the success rate of the blood samples between groups | after procedure
  if the blood sample will be succeeded: success , if the blood sample is failed : failure
Evaluate the impact of anxiety on the pain experienced just before the procedure | just before procedure
  anxiety will be measured with the STAI-Y just before the procedure
Time taken to perform the arterial puncture | start and end time of the arterial puncture
  the time of the blood sample will be noted
Compare patient satisfaction or perception of the procedure between groups | end of procedure
  the satisfaction will be assessed with likert scale ("Are you satisfied with the care you received during the blood gas analysis?: Strongly agree, Agree, Neither agree nor disagree, Disagree, Strongly disagree)

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU Brest, Brest, Finistere
  - CH Morlaix, Morlaix, Finistere

IPD SHARING:
Plan to Share IPD: Undecided